CLINICAL TRIAL: NCT04413994
Title: Effects of an Exclusive Human-milk Diet in Preterm NEOnates on Early VASCular Aging Risk Factors (NEOVASC)
Brief Title: Exclusive Human-milk in Preterm NEOnates and Early VASCular Aging Risk Factors (NEOVASC)
Acronym: NEOVASC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prolacta Bioscience (Industry)
Collaborators: Medical University of Vienna (Other); Federal University Teaching Hospital, Feldkirch, Austria (Other); Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Ursula Kohlendorfer, Professor, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEOVASC; 868624 (Other Grant/Funding Number: Austrian Research Promotion Agency)
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Prematurity; Vascular Aging
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The NEO-VASC study is a multicentric, prospective, randomized, controlled, open and parallel group clinical trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Randomized study product group (Active Comparator): receiving study product (human milk fortifier "Humavant") until a gestational age of 36 weeks
  Interventions: Dietary Supplement: Humavant
- Randomized control group (Active Comparator): receiving study product until a gestational age of 32 weeks and reference product (bovine based fortifier or bovine formula) after 32 weeks of gestation
  Interventions: Dietary Supplement: Humavant
- Term control group (No Intervention): Term-born controls as a reference group for outcome parameters

INTERVENTIONS:
Dietary Supplement: Humavant — Premature infants are randomized to either:
  1. An exclusive human milk diet which contains mother's milk or pasteurized donor human milk and the human milk fortifier until 36 weeks of gestation; OR
  2. Human milk (as long as available) and the human milk fortifier (as long as human milk is available) until a maximum of 32 weeks of gestation and thereafter human milk with a bovine-based fortifier or preterm formula.
  After 36 weeks of gestation, human milk with a bovine-based fortifier or preterm formula is used in both groups. As a control group, term-born age-matched controls are included.
  Arms: Randomized control group; Randomized study product group

SUMMARY:
Early vascular aging has its origins in fetal and neonatal life. The NEOVASC clinical trial aims to determine the effects of an exclusive human milk diet in extremely preterm infants on long-term cardiovascular health.

DETAILED DESCRIPTION:
Early vascular aging has its origins in fetal and neonatal life. This early period of life plays an important role in the development of obesity, high blood pressure, abnormalities in lipid metabolism and non-insulin dependent diabetes. Increased cardiovascular risk in formerly preterm infants constitutes a health problem of steadily growing relevance. Emerging evidence suggests that human milk feeding has substantial benefits to the health of all infants, especially for those born prematurely. Unfortunately, human milk alone does not provide sufficient concentrations of nutrients, especially calcium, phosphorus, protein, and fat needed for these infants to grow satisfactorily. For that purpose, fortifiers are used to help increase the nutritional value of human milk.

The NEOVASC study is a multicentric, prospective, randomized, controlled, open and parallel group clinical trial. A total of 200 extremely preterm infants and 100 term infants are recruited for the test and control group, respectively. Infants in the test group (i.e., premature neonates) are randomized to either:

1. An exclusive human milk diet which contains mother's milk or pasteurized donor human milk and a human milk fortifier until 36 weeks of gestation; OR
2. Human milk (as long as available) and a human milk fortifier (as long as human milk is available) until a maximum of 32 weeks of gestation and thereafter human milk with a bovine-based fortifier or preterm formula.

After 36 weeks of gestation, human milk with a bovine-based fortifier or preterm formula is used in both groups. As a control group, term-born age-matched controls are included. Participants within this control group are not enrolled at the time of birth but instead recruited in various kindergartens at the age of five. Therefore, data from birth is taken from the mother-child-booklet, which contains clinical records about the pregnancy, birth and early life of children born in Austria. The total study duration is scheduled for 96 months with a recruitment phase of 36 months. Follow-up visits are planned at one, two and five years of age for the test group.

The purpose of the NEOVASC clinical trial is to characterize early life stressors by assessing the effects of a physiological (i.e., human milk-based) nutrition in extremely preterm infants during the vulnerable preterm period on the risk of metabolic and vascular complications in later life. Outcomes include predictors and intermediate components of cardiovascular disease.

ELIGIBILITY:
Preterm-born group:

Inclusion Criteria:

1. Extremely preterm infants with a birth weight of 500-1250g.
2. Feeding is NPO or exclusive human milk prior to enrollment.
3. Parent(s) willing to sign informed consent.-

Exclusion Criteria:

1. Infants with a birth weight <500g or >1250g
2. Subjects diagnosed with inborn errors of metabolism such as galactosemia, phenylketonuria
3. Subjects who have not been NPO or fed exclusive human milk diet prior to enrollment.
4. Presence of major congenital malformation.
5. Presence of intestinal perforation or Stage 2 Necrotizing enterocolitis prior to enrollment.
6. Parent(s) not willing to sign informed consent.
7. Unable to participate for any reason based on the decision of the study investigator (e.g. unlikely to survive the study period).

Term-born group:

Inclusion criteria

1. Term-born children with an adequate birth weight
2. Parent(s) willing to sign informed consent

Exclusion criteria

1. Subjects with acute or chronic illness
2. Parent(s) not willing to sign informed consent

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | "First day of life" up to "five years of life"
  Primary outcome is the difference in fasting blood glucose at five years of age
Blood pressure | "First day of life" up to "five years"
  Primary outcome is the difference in blood pressure at five years of age
Distensibility of aorta | "First day of life" up to "five years"
  Primary outcome is the difference in the distensibility of the descending aorta using validated echocardiographic protocols at five years of age

SECONDARY OUTCOMES:
Fasting blood glucose | "First day of life" up to "24 months"
  Secondary outcome is fasting glucose at a corrected age of one and two years.
Blood pressure | "First day of life" up to "24 months"
  Secondary outcome is blood pressure at a corrected age of one and two years.
BMI | "First day of life" up to "five years"
  Secondary outcome is BMI at five years of age, weight in kilograms and height in meters will be combined to report BMI in kg/m2
Insulin sensitivity | "First day of life" up to "five years"
  Secondary outcome is insulin sensitivity at five years of age
Lipid profile | "First day of life" up to "five years"
  Secondary outcome is lipid profile at five years of age

OTHER OUTCOMES:
Fasting blood glucose | "five years of age"
  Difference in fasting blood glucose between preterm- and term-born children at five years of age
Blood pressure | "five years of age"
  Difference in blood pressure between preterm- and term-born children at five years of age
Distensibility of the descending aorta | "five years of age"
  Difference in the distensibility of the descending aorta between preterm- and term-born children using validated echocardiographic protocols at five years of age Results will be compared to results of term-born children
BMI | "five years of age"
  Difference in BMI between preterm- and term-born children at five years of age, weight in kilograms and height in meters will be combined to report BMI in kg/m2
Insulin sensitivity | "five years of age"
  Difference in insulin sensitivity between preterm- and term-born children at five years of age
Lipid profile | "five years of age"
  Difference in lipid profile between preterm- and term-born children at five years of age

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Kiechl-Kohlendorfer, MD, MSc, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitterer W, Binder C, Blassnig-Ezeh A, Auer-Hackenberg L, Berger A, Simma B, Wald M, Lee M, Kiechl-Kohlendorfer U. Effects of an exclusive human-milk diet in preterm neonates on early vascular aging risk factors (NEOVASC): study protocol for a multicentric, prospective, randomized, controlled, open, and parallel group clinical trial. Trials. 2021 Jul 31;22(1):509. doi: 10.1186/s13063-021-05445-9. PMID 34332629